CLINICAL TRIAL: NCT00462137
Title: The Influence of Hypnotic Medications on Sleep Arousal and Its Effect on Gastroesophageal Reflux
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 06U.101
Record Dates: First submitted 2007-02-01; First posted 2007-04-18 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Gastroesphageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: control group
  Interventions: Procedure: Sleep Studies
- 2: hypnotic group
  Interventions: Procedure: Sleep Studies

INTERVENTIONS:
Procedure: Sleep Studies

SUMMARY:
This is a continuation of a study that has already been completed in the division of gastroenterology (GI) looking at the effects of sleep medication zolpidem (Ambien) on subjects with Gastroesophageal reflux disease (GERD). That study looked at 16 subjects, 8 who had been diagnosed with GERD and 8 who did not have GERD (IRB Control #04S.41). All subjects previously had a PH probe completed in the division of GI at Thomas Jefferson University. An additional 8 subjects with GERD will be recruited to obtain more data to add to the previous study results. These subjects will undergo 2 sleep studies, one in which they will be given Ambien and one in which they will not.

DETAILED DESCRIPTION:
The use of hypnotic medications for the treatment of insomnia has increased as has the incidence of gastroesophageal reflux disease (GERD) and its complications. Nocturnal acid reflux is associated with severe injuries such as narrowing of the esophagus, inflammation and cancer of the esophagus.

A Gallup survey conducted in 2000, on behalf of the American Gastroenterological Association, found that 79% of respondents reported heartburn at night and 75% reported that symptoms affected their sleep. The impact that hypnotic medications (sleep medications) have on nocturnal reflux has not been well established. Orr et al. demonstrated that sleep arousal is critical in clearing acid from the esophagus and that decreased wakefulness results in prolonged esophageal acid exposure. Singh et al. showed that use of the hypnotic alprazolam, increases esophageal acid exposure time, possibly by blunting arousal and thereby interfering with acid clearance mechanisms. No study has examined sleep architecture and pattern (i.e. polysomnography) with and without hypnotic medication use and correlated this with how long the esophagus is exposed to acid.

Esophageal motility, gravity and salivation are three primary mechanisms by which acid is removed from the esophagus. Blunting nocturnal arousal with hypnotic medications may exacerbate gastroesophageal reflux or trigger it in otherwise healthy subjects, independent of any effects the medication may have on lower esophageal sphincter pressure. By depressing consciousness with pharmacologic agents (i.e. hypnotics, anxiolytics, antipsychotics) the body's defense against esophageal acid clearance may be impaired. Primary peristalsis, salivation and the warning symptoms of GERD are lost, thereby exposing the esophagus to a greater number and duration of GERD events.

The potential deleterious effects that hypnotic medications may have on nocturnal GERD has important implications on understanding the impact that hypnotic medications have on GERD.

The aim of this pilot study is to evaluate the effect that zolpidem (Ambien) has on sleep pattern, nocturnal GERD and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have had a pH probe test at Thomas Jefferson University between July 2004 and January 2006 with findings consistent with GERD.
* Male or female over the age of 18

Exclusion Criteria:

* Hypersensitivity to zolpidem or any of its components
* Pregnancy
* History of depression or hypnotic/substance abuse
* Prior esophagus or stomach surgery
* GI tract motility disorder
* Any sleep disorder or contraindications to the use of hypnotic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who have esophageal reflux
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Do hypnotic medications effect sleep arousal due to gi reflux? | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J DiMArino, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States